CLINICAL TRIAL: NCT03013998
Title: A Master Protocol for Biomarker-Based Treatment of AML (The Beat AML Trial)
Brief Title: Study of Biomarker-Based Treatment of Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beat AML, LLC (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BAML-16-001
Record Dates: First submitted 2016-12-21; First posted 2017-01-09 (Estimated); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Previously Untreated Relapsed Refractory Acute Myeloid Leukemia
Keywords: SNDX-5613; ZE46-0134; Ficlatuzumab; Revumenib; Lomonitinib
MeSH Terms: interventions — samalizumab; BI 836858; Daunorubicin; Cytarabine; Azacitidine; enasidenib; 6-(1H-indazol-6-yl)-N-(4-morpholinophenyl)imidazo(1,2-a)pyrazin-8-amine; Decitabine; pevonedistat; ivosidenib; gilteritinib; AZD5153; venetoclax; dubermatinib; AZD5991; ficlatuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (18):
- BAML-16-001-S17 (Experimental): This is an open-label Phase 1b dose escalation and expansion clinical trial to determine the safety and recommended dose of SNDX-5613 combined with azacitidine and venetoclax in newly diagnosed, untreated AML patients age ≥ 60 years who are not candidates or do not wish to pursue intensive induction therapy and who have NPM1 mutated or MLL-rearranged disease. After determination of the recommended dose of SNDX-5613, the study will have an expansion cohort to be treated at the recommended dose in combination with azacitidine and venetoclax in the same patient population.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: SNDX-5613 (BAML-16-001-S17); Drug: Azacitidine (BAML-16-001-S17); Drug: Venetoclax (BAML-16-001-S17)
- BAML-16-001-S12 (Arm A) (Active Comparator): This is an open label phase 2 randomized study in which eligible AML patients will be randomly assigned (1:1) to receive either the FDA label-approved regimen of 28-day Venetoclax + Azacitidine (Arm A) or the 14-day regimen of Venetoclax + Azacitidine (Arm B). Newly diagnosed acute myeloid leukemia (AML) patients ≥ 60 years will be enrolled.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Venetoclax (BAML-16-001-S12 Arm A); Drug: Azacitidine (BAML-16-001-S12 Arm A)
- BAML-16-001-S12 (Arm B) (Experimental): This is an open label phase 2 randomized study in which eligible AML patients will be randomly assigned (1:1) to receive either the FDA label-approved regimen of 28-day Venetoclax + Azacitidine (Arm A) or the 14-day regimen of Venetoclax + Azacitidine (Arm B). Newly diagnosed acute myeloid leukemia (AML) patients ≥ 60 years will be enrolled.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Venetoclax (BAML-16-001-S12 Arm B); Drug: Azacitidine (BAML-16-001-S12 Arm B)
- BAML-16-001-S21 (Group 1) (Experimental): This is a Phase 1, open-label, multicenter, dose escalation, and dose optimization study to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and preliminary efficacy of ZE46-0134 in adult patients with relapsed or refractory AML with FLT3-ITD and/or FLT3-TKD mutations for Group 1 and with spliceosome (SF3B1, SRSF2, U2AFI and ZRSR2) mutations for Group 2. Patients with AML that are out-patients or hospitalized due to their AML can be enrolled in the study. The study will be run in 2 parts: Part 1 will be dose escalation and determination of the maximum tolerated dose, and Part 2 will be dose expansion.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: ZE46-0134 (BAML-16-001-S21 Group 1)
- BAML-16-001-S21 (Group 2) (Experimental): This is a Phase 1, open-label, multicenter, dose escalation, and dose optimization study to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and preliminary efficacy of ZE46-0134 in adult patients with relapsed or refractory AML with FLT3-ITD and/or FLT3-TKD mutations for Group 1 and with spliceosome (SF3B1, SRSF2, U2AFI and ZRSR2) mutations for Group 2. Patients with AML that are out-patients or hospitalized due to their AML can be enrolled in the study. The study will be run in 2 parts: Part 1 will be dose escalation and determination of the maximum tolerated dose, and Part 2 will be dose expansion.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: ZE46-0134 (BAML-16-001-S21 Group 2)
- BAML-16-001-S24 (Experimental): This is a multi-center open-label Phase 1b safety run-in study followed by a Phase 2 study of ficlatuzumab given in combination with venetoclax azacitidine, in newly diagnosed untreated acute myeloid leukemia age ≥ 60 years who are not candidates or do not wish to pursue intensive induction therapy.
  Interventions: Drug: ficlatuzumab (BAML-16-001-S24); Drug: Azacitidine (BAML-16-001-S24); Drug: Venetoclax (BAML-16-001-S24)
- BAML-16-001-S1 (Closed) (Experimental): This is an open-label Phase 1b/2 clinical study of Samalizumab given in addition to standard induction chemotherapy/consolidation, followed by Samalizumab maintenance, in newly diagnosed acute myeloid leukemia. Patients that are marker negative, as defined based on the Beat AML Master Protocol assignment or with CBF karyotype/interphase cytogenetics/molecular testing defined by presence of t(8;21)(q22;q22) or the molecular equivalent RUNX1/RUNX1T1 fusion transcript or inv(16)(p13q22) or t(16;16)(p13;q22) or the molecular equivalent CBFB/MYH11 fusion transcript based on the Beat AML will receive Samalizumab in combination with induction therapy followed by Samalizumab maintenance.
  Interventions: Biological: Samalizumab (BAML-16-001-S1); Drug: Daunorubicin (BAML-16-001-S1); Drug: Cytarabine (BAML-16-001-S1)
- BAML-16-001-S2 (Closed) (Experimental): This is an open-label Phase 1b/2 clinical study of BI 836858 given in combination with azacitidine, followed by BI 836858 plus azacitidine maintenance, in newly diagnosed acute myeloid leukemia. The target population is assigned by the Beat AML Master Protocol (the "umbrella" study). Eligible patients will have previously untreated acute myeloid leukemia, age greater than or equal to 60, with any 1 of the following: mutated TET2, IDH1, IDH2, or WT1, or "marker negative" as defined by the overall Beat AML umbrella protocol.
  Interventions: Biological: BI 836858 (BAML-16-001-S2); Drug: Azacitidine (BAML-16-001-S2)
- BAML-16-001-S3 (Closed) (Experimental): This is a phase 2 clinical trial to assess the feasibility and efficacy of a stepwise approach to the treatment of IDH2-mutant AML. On day 1 of the trial, all enrolled participants will be initiated on therapy with the IDH2 inhibitor AG-221 for IDH2 R140 and R172-mutant patients. The dosing will be based on phase 1 experience of AG-221, which has established 100 mg daily as a safe and tolerated dose, with preliminary suggestion of efficacy. These will be administered continuously in 28 day cycles. Hydroxyurea will be allowed for the purposes of cytoreduction.
  Interventions: Drug: AG-221 (BAML-16-001-S3); Drug: Azacitidine (BAML-16-001-S3)
- BAML-16-001-S4 (Closed) (Experimental): This is a 2 cohort phase 1b/2 clinical trial to assess the feasibility and efficacy of entospletinib (ENTO) stepwise approach to the treatment of patients with balanced translocations of MLL identified cytogenetically (Cohort 1) and patients with MLL-partial tandem duplications identified molecularly (Cohort 2). All enrolled participants will be initiated on monotherapy with ENTO 400 mg PO BID. This dose will be administered continuously in 28 day cycles.
  Interventions: Drug: Entospletinib (BAML-16-001-S4); Drug: Azacitidine (BAML-16-001-S4)
- BAML-16-001-S5 (Closed) (Experimental): This is a phase 2 clinical trial to assess the feasibility and efficacy of a stepwise approach to the treatment of patients with TP53 mutations (identified molecularly) with/without complex karyotype (Cohort A) or complex karyotype (3 or greater metaphase abnormalities without TP53) (Cohort B). All enrolled participants will be initiated on entospletinib 400 mg orally twice daily. This dose will be administered continuously in 28 day cycles.
  Interventions: Drug: Entospletinib (BAML-16-001-S5); Drug: Decitabine (BAML-16-001-S5)
- BAML-16-001-S6 (Closed) (Experimental): The study is an open-label phase 2 study of entospletinib in younger and older AML patients with NPM1+/FLT3ITD-AML. It includes patients age ≥18 years who are able and willing to receive 7 + 3 intensive chemotherapy. Entospletinib is administered daily with IV daunorubicin (days 1-3 for Cycle 1) and cytarabine (days 1-7 for Cycle 1). If a second induction is required, it is given with IV daunorubicin (days 1-2 for Cycle 2) and cytarabine (days 1-5 for Cycle 2).
  Interventions: Drug: Entospletinib (BAML-16-001-S6); Drug: Daunorubicin (BAML-16-001-S6); Drug: Cytarabine (BAML-16-001-S6)
- BAML-16-001-S8 (Closed) (Experimental): This is an open-label Phase 1b/2 clinical study of gilteritinib monotherapy, gilteritinib in combination with decitabine, or gilteritinib in combination with decitabine and venetoclax in untreated FLT3 mutated AML with high and low variant allele frequency. Initially, the combination of gilteritinib and decitabine was tested (Group 1); however, subsequently the combination of decitabine and venetoclax was shown to be a highly effective therapy for older AML patients, so the triple combination of gilteritinib in combination with decitabine and venetoclax (Group 2) is now being evaluated in this study.
  Interventions: Drug: Gilteritinib (BAML-16-001-S8 Group 1); Drug: Decitabine (BAML-16-001-S8 Group 1); Drug: Decitabine (BAML-16-001-S8 Group 2); Drug: Venetoclax (BAML-16-001-S8 Group 2); Drug: Gilteritinib (BAML-16-001-S8 Group 2)
- BAML-16-001-S9 (Closed) (Experimental): This is an open-label phase 2 clinical trial of a stepwise approach to the treatment of patients with TP53 mutation AML. On day 1, all enrolled participants will be initiated on therapy with pevonedistat (20 mg/m2) day 1, 3 and 5 together with azacitidine (75 mg/m2 days 1-7 or day 1-5 then day 8, 9) every 28 days. During cycle 1, patients with rapidly progressive disease or severe organ dysfunction, not correctable by hydroxyurea cytoreduction will not be eligible to continue. Those patients who achieved a response, defined as complete response or complete response with incomplete blood count recovery, by the end of cycle 4 will continue on pevonedistat and azacitidine until disease progression, unacceptable toxicity, or 12 cycles of therapy. After 12 months of combined therapy, pevonedistat will be continued until progression of disease, unacceptable toxicity, or up to 2 years of total therapy.
  Interventions: Drug: Pevonedistat (BAML-16-001-S9); Drug: Azacitidine (BAML-16-001-S9)
- BAML-16-001-S10 (Closed) (Experimental): This is a phase 1b/2 clinical trial to assess the safety and efficacy of the combination of AZD5153 and venetoclax. In a phase 1b component, safety and tolerability of the combination will be assessed in relapsed/refractory AML patients ≥ 18 years of age. Following determination of the recommended Phase 2 dose (RP2D), newly diagnosed, marker negative patients age ≥ 60 will be enrolled in the phase 2 component; these patients will be treated at the previously identified RP2D for the combination. The RP2D will be the highest dose level with ≤ 1 out of 6 patients with dose limiting toxicity and defined as the maximum tolerated dose.
  Interventions: Drug: AZD5153 (BAML-16-001-S10); Drug: Venetoclax (BAML-16-001-S10)
- BAML-16-001-S14 (Closed) (Experimental): The study is an open-label Phase 1b/2 clinical study of TP-0903 given in addition to decitabine in patients ≥ 60 years with newly diagnosed, previously untreated AML with TP53 mutations and/or complex karyotype. The Phase 1b portion of this study will use a standard 3 + 3 design with dose escalation based upon dose limiting toxicities. The maximum tolerated dose will be defined as the highest dose where at most 1 patient in 6 experiences dose-limiting toxicity, and this is generally the recommended Phase 2 dose (RP2D). Once the RP2D is determined from Phase 1b, patients will be enrolled at this dose level to initiate the Phase 2 portion of the study.
  Interventions: Drug: TP-0903 (BAML-16-001-S14); Drug: Decitabine (BAML-16-001-S14)
- BAML-16-001-S16 (Closed) (Experimental): This is an open-label phase 2 clinical study to assess the feasibility and efficacy of a combination based approach to the treatment of IDH1 mutant AML. On day 1 of the trial, all enrolled participants will be initiated on therapy with the IDH1 inhibitor AG-120 given daily together with azacitidine (days 1-5 and 8-9 or 7 consecutive days 1-7) in 28 day cycles for IDH1 mutant patients. Those patients who have achieved a response, defined as complete response or complete response with incomplete blood count recovery, by the end of cycle 6, will continue on combination therapy for a total of 12 cycles and then patients will go onto receive monotherapy with AG-120 until disease progression or unacceptable side effects that mandate discontinuation of therapy. Patients who cannot complete 12 cycles of azacitidine may proceed onto monotherapy with AG-120.
  Interventions: Drug: AG-120 (BAML-16-001-S16); Drug: Azacitidine (BAML-16-001-S16)
- BAML-16-001-S18 (Closed) (Experimental): This is an open-label Phase 1b clinical study of AZD5991 + azacitidine in patients aged ≥60 years with newly diagnosed, previously untreated, hypermethylated and marker-negative AML. The phase 1b1 study will adopt a standard 3+3 design with dose escalation based upon dose limiting toxicities. The recommended Phase 2 dose (RP2D) is defined in this study as the highest dose level where less than 2 dose limiting toxicities (DLT) are observed out of 6 patients. Once the RP2D is defined, patients will be enrolled into 2 separate cohorts (hypermethylation and marker negative group) for the phase 1b2 expansion. These 2 groups will both be treated at the RP2D determined from phase 1b1.
  Interventions: Drug: AZD5991 (BAML-16-001-S18); Drug: Azacitidine (BAML-16-001-S18)

INTERVENTIONS:
Biological: Samalizumab (BAML-16-001-S1) — 300 mg/m2, IV, on days 1, 3, and 24; followed by 300 mg/m2, IV, every 21 days for 2 years in the absence of toxicity or disease progression. Dose may be de-escalated to 150 mg/m2 or escalated to 600 mg/m2 based on occurrence of dose-limiting toxicity.
  Arms: BAML-16-001-S1 (Closed)
Biological: BI 836858 (BAML-16-001-S2) — 20 mg/m2, IV, on days 9, 16, and 23 of a 28-day cycle; followed 20 by mg/m2, IV, on days 1, 8, 15 and 22 of each 28-day cycle for 2 years in the absence of toxicity or disease progression (reduced to monthly administration in event of complete response or complete response with incomplete blood count recovery). Dose may be escalated to a maximum dose of 320 mg/m2 or de-escalated to 10 mg/m2 based on occurrence of dose-limiting toxicity.
  Arms: BAML-16-001-S2 (Closed)
Other: Laboratory Biomarker Analysis — Molecular genomic assessment to assign patients to targeted therapy (sub-study) based on their specific subtype of acute myeloid leukemia
  Arms: BAML-16-001-S12 (Arm A); BAML-16-001-S12 (Arm B); BAML-16-001-S17; BAML-16-001-S21 (Group 1); BAML-16-001-S21 (Group 2)
Drug: Daunorubicin (BAML-16-001-S1) — 60 mg/m2, IV, on days 4, 5, and 6 of the induction cycle
  Arms: BAML-16-001-S1 (Closed)
Drug: Cytarabine (BAML-16-001-S1) — 100 mg/m2, IV, on days 4 through 10 of the 24-day induction cycle; 1000 mg/m2, IV, on days 2, 4, and 6 of the consolidation cycle 1 and days 1, 3, and 5 of consolidation cycles 2 through 4
  Arms: BAML-16-001-S1 (Closed)
Drug: Azacitidine (BAML-16-001-S2) — 75 mg/m2, IV, on days 1 through 7 of each 28-day cycle for 2 years in the absence of toxicity or disease progression
  Arms: BAML-16-001-S2 (Closed)
Drug: AG-221 (BAML-16-001-S3) — 100 mg, oral, daily until time of intolerance or disease progression. Dose may be de-escalated to 50 mg based on occurrence of dose-limiting toxicity.
  Other Names: Enasidenib
  Arms: BAML-16-001-S3 (Closed)
Drug: Azacitidine (BAML-16-001-S3) — 75 mg/m2, IV or SC, on days 1 through 7 of each 28-day cycle starting with cycle 6 and ending after 12 cycles for patients not attaining complete remission or complete remission with incomplete blood count recovery after 5 cycles of monotherapy with AG-221
  Arms: BAML-16-001-S3 (Closed)
Drug: Entospletinib (BAML-16-001-S4) — 200 mg, oral, twice daily for 5 years until time of intolerance or disease progression. Dose may be escalated to 400 mg.
  Other Names: GS-9973, ENTO
  Arms: BAML-16-001-S4 (Closed)
Drug: Azacitidine (BAML-16-001-S4) — 75 mg/m2, IV or SC, on days 1 through 7 of each 28-day cycle and continuing for 12 cycles. Treatment starts after 1 cycle of monotherapy with entospletinib for patients not attaining complete remission or complete remission with incomplete blood count recovery or after later cycles of monotherapy with entospletinib for patients with disease progression.
  Arms: BAML-16-001-S4 (Closed)
Drug: Entospletinib (BAML-16-001-S5) — 400 mg, oral, twice daily for 2 years on study until time of intolerance or disease progression. Dose may be de-escalated to 200 mg twice daily or 200 mg once daily based on occurrence of dose-limiting toxicity.
  Other Names: GS-9973, ENTO
  Arms: BAML-16-001-S5 (Closed)
Drug: Decitabine (BAML-16-001-S5) — 20 mg/m2, IV, on days 1 through 5 or 10 of each 28-day cycle and continuing for up to 11 cycles. During the first induction cycle, and the 2nd and 3rd induction cycles if they are needed, administration occurs on days 1 through 10 of each 28-day cycle. During subsequent consolidation, decitabine is administered on days 1 through 5 of each 28-day cycle and continuing for up to 11 cycles. Duration may be reduced by 1 day based on occurrence of dose-limiting toxicity, and patients may switch to entospletinib monotherapy maintenance at any time if they develop toxicity or are unwilling to continue decitabine during consolidation therapy.
  Arms: BAML-16-001-S5 (Closed)
Drug: Entospletinib (BAML-16-001-S6) — 400 mg, oral, twice daily for 2 years until time of intolerance or disease progression.
  Other Names: GS-9973, ENTO
  Arms: BAML-16-001-S6 (Closed)
Drug: Daunorubicin (BAML-16-001-S6) — 60 mg/m2, IV, on days 1-3 or 1-2 of each 28-day cycle for the first and second induction cycle, respectively
  Arms: BAML-16-001-S6 (Closed)
Drug: Cytarabine (BAML-16-001-S6) — 100 mg/m2, IV, on days 1 through 7 or 1 through 5 of each 28-day cycle for the first and second induction cycle, respectively; then 1000 mg/m2 (patients ≥60 years) or 3000 mg/m2 (younger patients with creatinine clearance >30 mL/min and <50 mL/min), IV, every 12 hours on days 1, 3, and 5 of each 28-day cycle for up to 4 consolidation cycles
  Arms: BAML-16-001-S6 (Closed)
Drug: Pevonedistat (BAML-16-001-S9) — 20 mg/m2, IV, on days 1, 3, and 5 of each 28-day cycle and continuing for 24 cycles in the absence of toxicity or disease progression
  Other Names: TAK-924, MLN4924
  Arms: BAML-16-001-S9 (Closed)
Drug: Azacitidine (BAML-16-001-S9) — 75 mg/m2, IV or SC, on days 1 through 7 or days 1 through 5 and then 8 through 9 (based on institutional guidelines) of each 28-day cycle and continuing for 12 cycles in the absence of toxicity or disease progression
  Arms: BAML-16-001-S9 (Closed)
Drug: AG-120 (BAML-16-001-S16) — 500 mg, oral, daily until time of intolerance or disease progression. Dose may be de-escalated to 250 mg based on occurrence of dose-limiting toxicity.
  Arms: BAML-16-001-S16 (Closed)
Drug: Azacitidine (BAML-16-001-S16) — 75 mg/m2, IV or SC, on days 1 through 7 or days 1 through 5 and then 8 through 9 (based on institutional guidelines) of each 28-day cycle and continuing for 12 cycles in the absence of toxicity or disease progression
  Arms: BAML-16-001-S16 (Closed)
Drug: Gilteritinib (BAML-16-001-S8 Group 1) — 120 mg, oral, daily, with treatment continuing based on bone marrow results at 28 and 56 days. Patients with partial response at 28 days continue treatment for an additional 28 days. Patients with complete remission (CR) or complete remission with incomplete hematologic recovery (CRi) at 28 or 56 days continue treatment for 5 years until time of intolerance or disease progression. Patients with less than partial response at 28 days or partial response at 28 days followed by less than CR or CRi at 56 days proceed to combination treatment with decitabine or non-study alternative.
  The combination dose is 80 mg, oral, daily, for 5 years until time of intolerance or disease progression (patients who do not achieve CR or CRi after 3 cycles will discontinue study treatment). The combination dose may be escalated to 120 mg daily or de-escalated to 80 mg daily given after decitabine rather than in combination with decitabine based on absence or occurrence of dose-limiting toxicity.
  Arms: BAML-16-001-S8 (Closed)
Drug: Decitabine (BAML-16-001-S8 Group 1) — 20 mg/m2, IV, on days 1 through 10 of each 28-day cycle and continuing for up to 3 cycles. Treatment starts after 1-2 cycles of monotherapy with gilteritinib if patients do not attain complete remission (CR) or complete remission with incomplete hematologic recovery (CRi) with monotherapy. Patients who do not achieve CR/CRi after 3 cycles of combination therapy will discontinue study treatment. If CR or CRi is obtained with combination therapy after 3 cycles, decitabine will be administered on days 1-5 of each subsequent 28-day cycle until progression, intolerance, or patient desire to discontinue therapy.
  Arms: BAML-16-001-S8 (Closed)
Drug: AZD5153 (BAML-16-001-S10) — 20 mg, oral, once daily during 7-day lead-in and then on days 1 through 21 of each 28-day cycle for up to 2 years or until allogeneic stem cell transplantation, time of intolerance, or disease progression [if the continuous administration AZD5153 on Days 1-21 of a 28-day cycle is not tolerated, an alternative schedule of 2 weeks on and 2 weeks off (i.e. AZD5153 will be administered on Days 1-14 of a 28-day cycle) will be explored]. Dose may be de-escalated to 10 mg or escalated to 30 mg based on occurrence of dose-limiting toxicity during phase 1 dose escalation. Starting with Cycle 2, patients may receive concomitant fluconazole, isavuconazole, or posaconazole and doses adjusted to 2, 5, or 8 mg daily. The Phase 1b expansion pharmacokinetics cohort will allow for posaconazole starting at Cycle 1 with AZD5153 dose adjusted from 10, 20, or 30 mg daily to 2, 5, or 8 mg daily. Phase 2 dose will be based on Phase 1 results.
  Arms: BAML-16-001-S10 (Closed)
Drug: Venetoclax (BAML-16-001-S10) — 400 mg, oral, on days 1 through 21 of each 28-day cycle and continuing for up to 12 cycles (for Cycle 1, day 1 dose will be 100 mg, day 2 dose 200 mg, and days 3 onward 400 mg). Starting with Cycle 2, patients may receive concomitant fluconazole or isavuconazole and daily doses adjusted to 200 mg, or posaconazole and daily doses adjusted to 70 mg. The Phase 1b expansion pharmacokinetics cohort will allow for posaconazole starting at Cycle 1 with Venetoclax dose adjusted to 10 mg on day 1, 20 mg on day 2, 50 mg on day 3, and 70 mg on day 4 onward).
  Arms: BAML-16-001-S10 (Closed)
Drug: TP-0903 (BAML-16-001-S14) — 37 mg, oral, once daily on days 1 through 21 of each 28-day cycle for up to 2 years to time of intolerance or disease progression. Dose may be de-escalated to as low as 12 mg or escalated to 50 mg based on occurrence of dose-limiting toxicity during Phase 1 dose escalation. Phase 2 dose will be based on Phase 1 results.
  Arms: BAML-16-001-S14 (Closed)
Drug: Decitabine (BAML-16-001-S14) — 20 mg/m2, IV, on days 1 through 5 or 10 of each 28-day cycle and continuing for up to 2 years to time of intolerance or disease progression. During the first induction cycle, and the 2nd and 3rd induction cycles if they are needed, administration occurs on days 1 through 10 of each 28-day cycle. During maintenance, decitabine is administered on days 1 through 5 of each 28-day cycle. Patients may switch to TP-0903 monotherapy maintenance if they develop toxicity or are unwilling to continue decitabine during maintenance therapy.
  Arms: BAML-16-001-S14 (Closed)
Drug: Decitabine (BAML-16-001-S8 Group 2) — 20 mg/m2, IV, on days 8 through 12 of the first 35-day induction cycle, then on days 1 through 5 of subsequent 28-day cycles and continuing for up to 60 cycles, disease progression, intolerance, or patient desire to discontinue therapy.
  Arms: BAML-16-001-S8 (Closed)
Drug: Venetoclax (BAML-16-001-S8 Group 2) — Oral dosing based on concurrent antifungal use. Dose without use of concomitant antifungal is 400mg, dose if on posaconazole is 70mg, dose if on voriconazole is 100mg, and dose if on moderate CYP3A inhibitors (ie fluconazole, isavuconazole) is 200mg continuing for up to 12 total cycles. For the 35-day induction cycle 1, dosing is days 2 through 28. For the 28-day induction cycle 2, if needed, dosing is days 1 through 21. For the 28-day consolidation cycles, dosing is days 1-15.
  Arms: BAML-16-001-S8 (Closed)
Drug: AZD5991 (BAML-16-001-S18) — 150 mg, IV, on days 1, 4, 8, 11, 15, and 18 of three 28-day cycles; followed by 150 mg/m2, IV, on days 1, 4, 8, and 11 of twenty-one 28-day cycles; followed by 150 mg/m2 on days 1 and 4 of each 28-day cycle until time of progression, unacceptable toxicity, death, or 57 total cycles of treatment. Dose may be escalated to a maximum dose of 400 mg or de-escalated to 100 mg based on occurrence of dose-limiting toxicity.
  Arms: BAML-16-001-S18 (Closed)
Drug: Azacitidine (BAML-16-001-S18) — 75 mg/m2, IV or SC, on days 1-7 or days 1-5 and 8 and 9 or days 1-2 and 5-9 (based on institutional guidelines) of each 28-day cycle until time of progression, unacceptable toxicity, death, or 57 total cycles of treatment
  Arms: BAML-16-001-S18 (Closed)
Drug: SNDX-5613 (BAML-16-001-S17) — Patients starting induction with CYP3A4 inhibitors will be dosed at 113 mg capsule or 110 mg tablet, oral, every 12 hours on Day 1-28 of each 28-day cycle, until time of progression, unacceptable toxicity, or death. Dose may be escalated to a maximum dose of 163 mg capsule or 220 mg tablet on days 1-28 or de-escalated to 113 mg on days 1-21 based on occurrence of dose-limiting toxicity. Other possible dose escalation and de-escalation would be 163 mg on days 1-21, 75 mg on days 1-21 and 75 mg on days 1-28. Patients starting treatment without CYP3A4 inhibitors will be dosed at 276 mg capsule (270 mg tablet) or 226 mg capsule (220 mg tablet) oral, every 12 hours on Day 1-28 of each 28-day cycle.
  Following completion of induction, patients who do not require strong CYP3A4 inhibitor antifungals will have daily doses increased for doses in range of 113-226 mg capsules or 110-220 mg tablets (days 1-21 or days 1-28).
  Arms: BAML-16-001-S17
Drug: Azacitidine (BAML-16-001-S17) — 75 mg/m2, IV or SC, on days 1-7 (during induction cycle/cycles) or can use alternative scheduled on days 1-5 and 8 and 9 or days 1-2 and 5-9 (based on institutional guidelines) during continued therapy cycles of each 28-day cycle until time of progression, unacceptable toxicity, or death.
  Arms: BAML-16-001-S17
Drug: Venetoclax (BAML-16-001-S17) — For Cycle 1 induction, day 1 dose is 10 mg, day 2 dose 20 mg, day 3 dose is 50 mg, and day 4 onward dose is 100 mg or 70 mg depending on concomitant antifungal treatment. For Cycles 2 and 3 inductions, daily doses are 100 or 70 mg depending on concomitant antifungal treatment. During continued therapy cycles, if not on concomitant strong CYP3A4 inhibitor antifungals, 400 mg, oral, on days 1 through 28 or days 1 through 14 of each 28-day cycle until time of progression, unacceptable toxicity, or death (patients on moderate CYP3A4 inhibitor antifungals should receive 200 mg/day).
  Arms: BAML-16-001-S17
Drug: Gilteritinib (BAML-16-001-S8 Group 2) — Phase 1b induction: 80-120 mg, oral, daily for day 1 up to day 28 of the 35-day induction cycle 1; then 80-120 mg, oral, daily for day 1 up to day 28 of the 28-day induction cycle 2 (induction cycle 2 administered if needed after cycle 1 based on results bone marrow evaluation). Phase 1b consolidation: 80-120 mg, oral, daily for day 1 up to day 21 of the 28-day cycles, for a total of 12 total induction and consolidation cycles. Phase 1b induction and consolidation dose and duration may be escalated or de-escalated based on occurrence of dose-limiting toxicity. Phase 2 induction and consolidation dosage to be based on results of Phase 1b. Phase 1b and 2 maintenance: 120 mg, oral, daily for 28 days of the 28-day cycles until patient is minimal residual disease negative for FLT3 based on scheduled bone marrow biopsy, progression of disease, unacceptable toxicities, or desire to discontinue therapy.
  Arms: BAML-16-001-S8 (Closed)
Drug: Venetoclax (BAML-16-001-S12 Arm A) — 400 mg, oral, on days 1 through 28 of each 28-day cycle for up to 2 cycles or until unacceptable toxicity or death. For Cycle 1, day 1 dose is 100 mg, day 2 dose 200 mg, and day 3 onward dose is 400 mg. (Dose adjusted by anti-fungal agent use per the package insert.)
  Arms: BAML-16-001-S12 (Arm A)
Drug: Azacitidine (BAML-16-001-S12 Arm A) — 75 mg/m2, IV or SC, on days 1-7 or days 1-5 and 8 and 9 or days 1-2 and 5-9 (based on institutional guidelines) of each 28-day cycle for up to 2 cycles or until unacceptable toxicity or death.
  Arms: BAML-16-001-S12 (Arm A)
Drug: Venetoclax (BAML-16-001-S12 Arm B) — 400 mg, oral, on days 1 through 14 of each 14-day cycle for up to 2 cycles or until unacceptable toxicity or death. For Cycle 1, day 1 dose is 100 mg, day 2 dose 200 mg, and day 3 onward dose is 400 mg. (Dose adjusted by anti-fungal agent use per the package insert.)
  Arms: BAML-16-001-S12 (Arm B)
Drug: Azacitidine (BAML-16-001-S12 Arm B) — 75 mg/m2, IV or SC, on days 1-7 or days 1-5 and 8 and 9 or days 1-2 and 5-9 (based on institutional guidelines) of each 14-day cycle for up to 2 cycles or until unacceptable toxicity or death.
  Arms: BAML-16-001-S12 (Arm B)
Drug: ZE46-0134 (BAML-16-001-S21 Group 1) — 10 mg to 100 mg oral on Days 1-28 of each 28-day cycle for up to 24 cycles. On the first day of Cycle 1, a loading dose of 30 mg to 200 mg will be administered, after which the daily maintenance dose of 10 mg to 100 mg will be administered on days 2-28 of Cycle 1. Maintenance dose continues in subsequence cycles, for up to 24 cycles total.
  Arms: BAML-16-001-S21 (Group 1)
Drug: ficlatuzumab (BAML-16-001-S24) — 10, 15 or 20 mg/kg IV on days 1 and 15.
  Arms: BAML-16-001-S24
Drug: Azacitidine (BAML-16-001-S24) — 75 mg/m2, IV or SC, on days 3-9 (during induction cycle 1) or can use alternative scheduled on days 3-7 and 10 and 11 or days 3-4 and 7-11 (based on institutional guidelines) for 30 days of Induction Cycle 1. All other induction cycle or continued therapy cycles of each 28-day cycle will be days 1-7, days 1-5 and 8-9 or days 1-2 and 5-9 (based on institutional guidelines) until time of progression, unacceptable toxicity, or death.
  Arms: BAML-16-001-S24
Drug: Venetoclax (BAML-16-001-S24) — For Cycle 1 induction, day 3 dose is 100 mg, day 4 dose 200 mg, day 5 onward dose is 400 mg, depending on concomitant antifungal treatment. For Cycles 2 and 3 inductions, daily doses are 400mg or lower depending on concomitant antifungal treatment. During continued therapy cycles, if not on concomitant strong CYP3A4 inhibitor antifungals, 400 mg, oral, on days 1 through 14 of each 28-day cycle until time of progression, unacceptable toxicity, or death (patients on moderate CYP3A4 inhibitor antifungals should receive 200 mg/day).
  Arms: BAML-16-001-S24
Drug: ZE46-0134 (BAML-16-001-S21 Group 2) — 60 mg to 200 mg oral on Days 1-28 of each 28-day cycle for up to 24 cycles, for up to 24 cycles total.
  Arms: BAML-16-001-S21 (Group 2)

SUMMARY:
This screening and multi-sub-study Phase 1b/2 trial will establish a method for genomic screening followed by assigning and accruing simultaneously to a multi-study "Master Protocol (BAML-16-001-M1)." The specific subtype of acute myeloid leukemia will determine which sub-study, within this protocol, a participant will be assigned to evaluate investigational therapies or combinations with the ultimate goal of advancing new targeted therapies for approval. The study also includes a marker negative sub-study which will include all screened patients not eligible for any of the biomarker-driven sub-studies. Patients with myeloid malignancies [e.g. myelodysplastic syndrome (MDS) or other diseases], will be allowed to enroll to Master protocol if there is an available sub-study.

ELIGIBILITY:
Inclusion Criteria:

* Adults, age 60 years or older at the time of diagnosis unless in a specific known cytogenetic and genomic group for which treatment in Group A, B, or C is allowed by the sub-study where age 18 and older is allowed. In such case, waiting for Foundation Medicine test results would not be required to proceed with sub-study treatment. Patients < 60 years old who are screened but do not fall within the cytogenetic and genomic open sub-studies would still be followed on the M1 Master Protocol and not considered screen fails.
* Patients must be able to understand and provide written informed consent
* Cohort Inclusion Criteria - Group A: Patients must have previously untreated acute myeloid leukemia (AML) according to the WHO classification with no prior treatment other than hydroxyurea. Patients with myeloid malignancies [e.g. myelodysplastic syndrome (MDS) or other disease], will be allowed to enroll to this group. For previously untreated subjects with ≥ 20% blasts in bone marrow or blood only: Prior therapy for myelodysplastic syndrome (MDS), myeloproliferative syndromes (MPD), or aplastic anemia is permitted. For select group, patients who cannot wait or choose not to wait for results of genomic testing as specified in this protocol, will be allowed to enroll to select sub-studies that allow enrollment and treatment of all patients regardless of their genomic mutations or cytogenetics. For this group, patients will proceed to enroll to that select sub-study without waiting for results of genomic testing and genomic samples will be collected to be analyzed retrospectively after patients' enrollment.
* Cohort Inclusion Criteria - Group B: Patients must have relapsed or refractory AML according to the WHO classification. For study purposes, refractory AML is defined as failure to ever achieve a complete response (CR) or recurrence of AML within 6 months of achieving CR; relapsed AML is defined as all others with disease after prior remission. For select genomic aberrations specified in the sub-studies, patients ≥ 18 years of age may be allowed to enroll in this portion of the study. Patients with relapsed or refractory myeloid malignancies (e.g., MDS or other diseases) will be allowed to enroll to this group.
* Cohort Inclusion Criteria - Group C: For select sites which are not part of the Beat AML core sites. These sites will only participate in select sub-studies. Patients in this group will enroll under the Beat AML M1 Master protocol with the intent to enroll into these select sub-studies and following screening on Beat M1 Master protocol, they will come off M1 Master protocol.

Exclusion Criteria:

* Acute promyelocytic leukemia
* Clinically active central nervous system (CNS) involvement by AML. A patient may be considered eligible if CNS leukemia is showing response to treatment at study entry and should continue to receive intrathecal therapy as clinical indicated. Patients who require or are undergoing craniospinal irradiation of disease control would not be eligible for participation.
* Signs of leukostasis requiring urgent therapy
* Disseminated intravascular coagulopathy with active bleeding or signs of thrombosis
* Patients with psychological, familial, social, or geographic factors that otherwise preclude them from giving informed consent, following the protocol (including failure to collect genomics samples for screening), or potentially hamper compliance with study treatment and follow-up
* Any other significant medical condition, including psychiatric illness or laboratory abnormality, that would preclude the patient participating in the trial or would confound the interpretation of the results of the trial.

BAML-16-001-S17 - Inclusion Criteria:

1. Patients, age 60 years or older at the time of diagnosis with untreated AML according to the International Consensus Classification (ICC) 2022 guidelines, that have NPM1 mutated or MLL rearranged disease and who are not candidates for or do not wish to pursue intensive induction chemotherapy.
2. Patients must be able to understand and provide written informed consent.
3. Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2.
4. Aspartate aminotransferase (AST) < 5 x upper limit of normal (ULN), alanine aminotransferase (ALT) < 5 x ULN, and total bilirubin < 2 x ULN (except for patients with known or suspected Gilbert's syndrome and with direct bilirubin within normal range) for the local laboratory.
5. Adequate renal function as defined by calculated creatinine clearance ≥ 60 mL/min for the local laboratory.
6. Females must be non-child bearing, postmenopausal, surgically sterile or meet certain criteria if of childbearing potential. Males must adhere to criteria if with females of child bearing potentia
7. Patients must have previously untreated AML with no prior treatment other than hydroxyurea. No chemotherapy for AML outside of hydroxyurea for treatment of leukostasis or ATRA for initially suspected APL (that is ruled out) is allowed as well as one dose of intrathecal chemotherapy for suspected CNS involvement (that is ruled out) is allowed. Prior therapy for myelodysplastic syndrome is (MDS) allowed except for hypomethylating agents.
8. If the patient has co-morbid illness or malignancy, life expectancy attributed to this must be greater than 2 years.

BAML-16-001-S17 - Exclusion Criteria:

1. Isolated myeloid sarcoma (meaning, patients must have blood or marrow involvement with AML to enter the study).
2. Acute promyelocytic leukemia (FAB M3).
3. Favorable risk cytogenetics [Core Binding Factor (CBF) AML].
4. Active central nervous system (CNS) involvement by AML.
5. Signs of leukostasis requiring urgent therapy.
6. Patients with WBC ≥ 25,000/μl. (Patients must have WBC < 25,000/μl to begin therapy and Hydroxyurea may be used to obtain this level).
7. Patients willing and able to receive intensive induction chemotherapy.
8. Disseminated intravascular coagulopathy with active bleeding or signs of thrombosis.
9. Patients with psychological, familial, social, or geographic factors that otherwise preclude them from giving informed consent, following the protocol, or potentially hamper compliance with study treatment and follow-up.
10. Any other significant medical condition, including psychiatric illness or laboratory abnormality, that would preclude the patient participating in the trial or would confound the interpretation of the results of the trial.
11. Known active Human Immunodeficiency Virus (HIV), active hepatitis B or active hepatitis C infection.
12. Patients with the following will be excluded: uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, serious cardiac arrhythmia, myocardial infarction as presentation of AML, New York Heart Association (NYHA) Class III or IV heart failure, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Patients with medical comorbidities that will preclude safety evaluation of the combination should not be enrolled.
13. As infection is a common feature of AML, patients with active infection are permitted to enroll provided that the infection is under control. Patients with uncontrolled infection shall not be enrolled until infection is treated and brought under control.
14. Patients who have received an investigational agent (for any indication) within 5 half-lives of the agent and until toxicity from this has resolved to grade 1 or less; if the half-life of the agent is unknown, patients must wait 4 weeks prior to first dose of study treatment. An investigational agent is one for which there is no approved indication by the United States (US) FDA.
15. Patients with QTcF (Fridericia) > 450 ms for male patients and > 468 for female patients; patients with right, left, or partial bundle branch blocks or pacemaker that may confound interpretation of this reading are excluded from this provided they lack history of primary arrhythmic events and are cleared by cardiology for enrollment in the trial. Any factors that increase the risk of QTc prolongation or risk of arrhythmic event such as congenital long QT syndrome or family history of long QT syndrome.

BAML-16-001-S21 - Inclusion Criteria:

1. Written Informed Consent must be obtained from the patient prior to any study-related procedures (including withdrawal of prohibited medication, if applicable).
2. Patient is ≥18 years of age at the time of obtaining informed consent.
3. Patient is refractory to or relapsed after multiple AML therapies (with or without HSCT). and have exhausted all reasonable therapies expected to produce benefit unless the patient declines or is ineligible for these.
4. Group 1: Patient must have a confirmed FLT3-ITD or FLT3-TKD mutation by central laboratory testing. Group 2: Patient must have a documented SF3B1, SRSF2, U2AF1, or ZRSR2 pathogenic mutation by local lab sequencing.
5. For Group 1 only: Patients must have previously been treated with Gilteritinib with failure to stop disease progression, or not met the criteria for treatment with Gilteritinib in the opinion of the Investigator or chosen not to have treatment with Gilteritinib.
6. Patients have a life expectancy of at least 3 months in the opinion of the Investigator.
7. Patient has an Eastern Cooperative Oncology Group (ECOG) performance status ≤2.
8. Patient must meet the following criteria as indicated on the clinical laboratory tests:

   1. Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 × upper limit of normal (ULN).
   2. Serum total bilirubin ≤1.5 × ULN unless due to Gilbert's disease where a maximum total bilirubin level of 4.0 mg/dL is acceptable.
   3. Estimated glomerular filtration rate (eGFR) of > >40 mL/min as calculated by the Modification of Diet in Renal Disease equation.
9. Females must be non-child bearing, postmenopausal, surgically sterile or meet certain criteria if of childbearing potential.
10. Males must adhere to criteria if with females of child bearing potential

BAML-16-001-S21 - Exclusion Criteria:

1. Diagnosis of isolated myeloid sarcoma (meaning, patients must have blood or marrow involvement with AML).
2. Acute promyelocytic leukemia (FAB M3).
3. Active central nervous system (CNS) involvement by AML.
4. Clinical signs/symptoms of leukostasis requiring urgent therapy.
5. Known active infection with Human Immunodeficiency Virus (HIV), hepatitis B or hepatitis C. Patients with a history of positive serology for hepatitis B or C require a negative Polymerase chain reaction (PCR) test for virus to go onto therapy.
6. Disseminated intravascular coagulopathy with active, unmanageable bleeding or signs of thrombosis.
7. Patients who have received an investigational agent (for any indication) within 5 half-lives of the agent; if the half-life of the agent is unknown, patients must wait 1 week prior to first dose of study treatment. An investigational agent is one for which there is no approved indication by the local regulatory authority.
8. Systemic chemotherapy or radiation therapy within 1 week prior to starting protocol with the exception of hydroxyurea, which is allowed to control white blood cell counts.
9. Female patients who are pregnant or lactating.
10. Patients with QTcF > 470 msec that cannot be corrected with electrolyte replacement, hydration, or medication modifications.
11. Patients with psychological, familial, social, or geographic factors, other significant medical condition, laboratory abnormality that otherwise preclude them from giving informed consent, following the protocol, potentially hamper compliance with study treatment and follow-up or would confound the interpretation of the results of the study.
12. Patients with the following will be excluded: uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, serious cardiac arrhythmia, myocardial infarction with evidence of residual abnormalities within 6 months prior to enrollment (Troponin (regular or high sensitivity) leak alone not included if no residual dysfunction), New York Heart Association (NYHA) Class III or IV heart failure, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Patients with medical comorbidities that will preclude safety evaluation of the combination should not be enrolled.
13. Infection is a common feature of AML, as such patients with active infection are permitted to enroll provided that the infection is under control in the opinion of the Investigator. Patients with uncontrolled infection shall not be enrolled until infection is treated and brought under control.

BAML-16-001-S24 - Inclusion Criteria:

1. ≥ 60 years at time of AML diagnosis
2. Eastern Cooperative Oncology Group (ECOG) score of 0, 1, or 2
3. Aspartate aminotransferase (AST) < 2.5 x upper limit of normal (ULN), alanine aminotransferase (ALT) < 2.5 x ULN, and total bilirubin < 1.5 x ULN (except for patients with known Gilbert's syndrome) for the local laboratory. If due to disease, higher values may be approved after discussion with medical monitor.
4. Adequate renal function as defined by calculated creatinine clearance > 40 mL/min per the local laboratory
5. Patients must be able to understand and provide written informed consent.
6. Females must be non-child bearing, postmenopausal, surgically sterile or meet certain criteria if of childbearing potential.
7. Males must adhere to criteria if with females of child bearing potential
8. No prior chemotherapy for leukemia, except hydroxyurea to control leukocytosis and ATRA for initially suspected APL, which is permitted. [Prior therapy for myelodysplastic syndrome (MDS) or myeloproliferative neoplasm (MPN) allowed except for hypomethylating agents].
9. If the patient has co-morbid illness or malignancy, life expectancy attributed to this must be greater than 2 years.

BAML-16-001-S24 - Exclusion Criteria:

1. Patients able and willing to receive intensive induction chemotherapy for underlying AML.
2. Isolated myeloid sarcoma (meaning, patients must have blood or marrow involvement with AML to enter the study).
3. Acute promyelocytic leukemia.
4. Known active central nervous system (CNS) involvement by AML.
5. Clinical signs/symptoms of leukostasis requiring urgent therapy.
6. Known active Human Immunodeficiency Virus (HIV), active hepatitis B or active hepatitis C infection.
7. Disseminated intravascular coagulopathy with active bleeding or signs of thrombosis.
8. Patients who have received an investigational agent (for any indication) within 5 half-lives of the agent; if the half-life of the agent is unknown, patients must wait 1 week prior to first dose of study treatment. An investigational agent is one for which there is no approved indication by the United States (US) FDA.
9. Systemic antineoplastic therapy (for any indication) within 5 half-lives or radiation therapy within 1 week prior to starting protocol except for hydroxyurea, which is allowed to control white blood cell counts.
10. Patients with psychological, familial, social, or geographic factors, other significant medical condition, laboratory abnormality that otherwise preclude them from giving informed consent, following the protocol, potentially hamper compliance with study treatment and follow-up or would confound the interpretation of the results of the trial.
11. Patients with the following will be excluded: uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, serious cardiac arrhythmia, myocardial infarction within 6 months prior to enrollment (Troponin leak alone not included if no residual dysfunction) New York Heart Association (NYHA) Class III or IV heart failure, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Patients with medical comorbidities that will preclude safety evaluation of the combination should not be enrolled.
12. As infection is a common feature of AML, patients with active infection are permitted to enroll provided that the infection is under control. Patients with uncontrolled infection shall not be enrolled until infection is treated and brought under control.
13. Patients who require treatment with concomitant drugs that are strong inducers of cytochrome P450 (CYP) 3A.
14. Patients who require treatment with concomitant drugs that are strong inhibitors or inducers of P-glycoprotein (P-gp) with the exception of drugs that are considered absolutely essential for the care of the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2016-11; Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients for whom molecular, immunophenotypic, and/or biochemical studies are completed in < 7 calendar days for assignment of treatment | 7 days
  The feasibility of completing molecular, genetic, immunophenotypic, and biochemical testing for assignment of therapy will be assessed based on the proportion of patients for whom testing is completed within 7 days of the registration sample arriving at the laboratory
Proportion of patients assigned to a novel therapeutic treatment group in 1 of several sub-studies in this Master Protocol, based on the result of the molecular, immunophenotypic, and/or biochemical studies | 7 days
  The feasibility of assigning patients to a treatment group will be assessed based on the proportion who are eligible for screening in this study who are assigned to treatment either on this study or an industry study relevant to the specific marker group and not unassignable due to insufficient material, laboratory error, or any other factors
Clinical response rate (rate of complete and partial responses) according to International Working Group criteria for treatment outcomes in therapeutic trials in acute myeloid leukemia | Up to 5 years

SECONDARY OUTCOMES:
Proportion of patients enrolled on this trial that ultimately will be assigned and go onto an assigned therapy | 7 days
Dynamic changes in clonal architecture over time in acute myeloid leukemia patients receiving targeted therapies | time of diagnosis, remission (complete response or complete response with incomplete blood count recovery), 1 year of treatment, and relapse
Relationships between baseline functional status and response rate or progression-free survival based on graphical comparison (eg, side-by-side boxplots or Kaplan-Meier plots) | Up to 5 years
  Assessments of functional status will include Eastern Cooperative Oncology Group Performance Status. Assessment of clinical response will be made according to International Working Group criteria. Relationships will be explored graphically (eg, side-by-side boxplots or Kaplan-Meier plots), where estimates with confidence intervals will be presented as the primary method of analysis due to the limited number of patients.

CONTACTS AND LOCATIONS:
Overall Officials: John C Byrd, MD, Principal Investigator — Beat AML
Locations (19):
- United States (19):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - UCLA Ronald Reagan Medical Center, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - University of Colorado, Denver, Colorado
  - University of Florida Health Shands Cancer Hospital, Gainesville, Florida
  - Mayo Clinic Florida, Jacksonville, Florida
  - Emory University, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - University of Maryland Medical Center, Baltimore, Maryland
  - Mayo Clinic Minnesota, Rochester, Minnesota
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - UNC Hospitals, University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Ohio State University, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - University of Texas Southwestern, Dallas, Texas
  - Huntsman Cancer Institute, University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burd A, Levine RL, Ruppert AS, Mims AS, Borate U, Stein EM, Patel P, Baer MR, Stock W, Deininger M, Blum W, Schiller G, Olin R, Litzow M, Foran J, Lin TL, Ball B, Boyiadzis M, Traer E, Odenike O, Arellano M, Walker A, Duong VH, Kovacsovics T, Collins R, Shoben AB, Heerema NA, Foster MC, Vergilio JA, Brennan T, Vietz C, Severson E, Miller M, Rosenberg L, Marcus S, Yocum A, Chen T, Stefanos M, Druker B, Byrd JC. Precision medicine treatment in acute myeloid leukemia using prospective genomic profiling: feasibility and preliminary efficacy of the Beat AML Master Trial. Nat Med. 2020 Dec;26(12):1852-1858. doi: 10.1038/s41591-020-1089-8. Epub 2020 Oct 26. PMID 33106665
- [Background] Borate U, Yang F, Press R, Ruppert AS, Jones D, Caruthers S, Zhao W, Vergilio JA, Pavlick DC, Juckett L, Norris B, Bucy T, Burd A, Stein EM, Patel P, Baer MR, Stock W, Schiller G, Blum W, Kovacsovics T, Litzow M, Foran J, Heerema NA, Rosenberg L, Marcus S, Yocum A, Stefanos M, Druker B, Byrd JC, Levine RL, Mims A. Samples from patients with AML show high concordance in detection of mutations by NGS at local institutions vs central laboratories. Blood Adv. 2023 Oct 24;7(20):6048-6054. doi: 10.1182/bloodadvances.2022009008. PMID 37459200
- [Background] Rosenberg L, Levaux H, Levine RL, Shah A, Denmark J, Hereema N, Owen M, Kalk S, Kenny N, Vinson G, Vergilio JA, Mims A, Borate U, Blum W, Stein E, Gana TJ, Stefanos M, Yocum A, Marcus S, Shoben A, Druker B, Byrd J, Burd A. Streamlined Operational Approaches and Use of e-Technologies in Clinical Trials: Beat Acute Myeloid Leukemia Master Trial. Ther Innov Regul Sci. 2021 Sep;55(5):926-935. doi: 10.1007/s43441-021-00277-w. Epub 2021 May 16. PMID 33997942
- [Background] Cai SF, Huang Y, Lance JR, Mao HC, Dunbar AJ, McNulty SN, Druley T, Li Y, Baer MR, Stock W, Kovacsovics T, Blum WG, Schiller GJ, Olin RL, Foran JM, Litzow M, Lin T, Patel P, Foster MC, Boyiadzis M, Collins RH, Chervin J, Shoben A, Vergilio JA, Heerema NA, Rosenberg L, Chen TL, Yocum AO, Druggan F, Marcus S, Stefanos M, Druker BJ, Mims AS, Borate U, Burd A, Byrd JC, Levine RL, Stein EM. A study to assess the efficacy of enasidenib and risk-adapted addition of azacitidine in newly diagnosed IDH2-mutant AML. Blood Adv. 2024 Jan 23;8(2):429-440. doi: 10.1182/bloodadvances.2023010563. PMID 37871309
- [Background] Duong VH, Ruppert AS, Mims AS, Borate U, Stein EM, Baer MR, Stock W, Kovacsovics T, Blum W, Arellano ML, Schiller GJ, Olin RL, Foran JM, Litzow MR, Lin TL, Patel PA, Foster MC, Redner RL, Al-Mansour Z, Cogle CR, Swords RT, Collins RH, Vergilio JA, Heerema NA, Rosenberg L, Yocum AO, Marcus S, Chen T, Druggan F, Stefanos M, Gana TJ, Shoben AB, Druker BJ, Burd A, Byrd JC, Levine RL, Boyiadzis MM. Entospletinib with decitabine in acute myeloid leukemia with mutant TP53 or complex karyotype: A phase 2 substudy of the Beat AML Master Trial. Cancer. 2023 Aug 1;129(15):2308-2320. doi: 10.1002/cncr.34780. Epub 2023 Apr 20. PMID 37078412
- [Background] Saliba AN, Kaufmann SH, Stein EM, Patel PA, Baer MR, Stock W, Deininger M, Blum W, Schiller GJ, Olin RL, Litzow MR, Lin TL, Ball BJ, Boyiadzis MM, Traer E, Odenike O, Arellano ML, Walker A, Duong VH, Kovacsovics T, Collins RH, Shoben AB, Heerema NA, Foster MC, Peterson KL, Schneider PA, Martycz M, Gana TJ, Rosenberg L, Marcus S, Yocum AO, Chen T, Stefanos M, Mims AS, Borate U, Burd A, Druker BJ, Levine RL, Byrd JC, Foran JM. Pevonedistat with azacitidine in older patients with TP53-mutated AML: a phase 2 study with laboratory correlates. Blood Adv. 2023 Jun 13;7(11):2360-2363. doi: 10.1182/bloodadvances.2022008625. No abstract available. PMID 36315007
- [Derived] Eisenmann ED, Swords R, Huang Y, Orwick S, Buelow D, Abbott N, Phelps M, Zeidner J, Foster MC, Lin TL, Baer MR, Madanat YF, Kovacsovics T, Redner R, Al-Mansour Z, Bhatnagar B, Stefanos M, Martycz M, Druggan F, Chen TL, Yocum AO, Borate U, Druker BJ, Burd A, Levine RL, Byrd JC, Baker SD, Mims AS. A Phase 1b/2 Study of TP-0903 and Decitabine Targeting Mutant TP53 and/or Complex Karyotype in Patients with Untreated Acute Myeloid Leukemia >/=Age 60 Years. Cancer Res Commun. 2025 Jul 1;5(7):1129-1139. doi: 10.1158/2767-9764.CRC-25-0091. PMID 40557912
- [Derived] Zeidner JF, Lin TL, Welkie RL, Curran E, Koenig K, Stock W, Madanat YF, Swords R, Baer MR, Blum W, Stein EM, Olin RL, Schiller G, Nichols A, Odenike O, Traer E, Lachowiez C, Duong VH, Hochman MJ, Cai SF, Smith C, Stefanos M, Martycz M, Huang Y, Rosenberg L, Marcus S, Chen TL, Yocum AO, Druker BJ, Levine RL, Borate U, Byrd JC, Mims AS. Azacitidine, Venetoclax, and Revumenib for Newly Diagnosed NPM1-Mutated or KMT2A-Rearranged AML. J Clin Oncol. 2025 Aug 10;43(23):2606-2615. doi: 10.1200/JCO-25-00914. Epub 2025 Jun 12. PMID 40504618
- See also: Click here for more information about this study: Study of Biomarker-Based Treatment of Acute Myeloid Leukemia — https://www.BloodCancerUnited.org/beataml